CLINICAL TRIAL: NCT03456414
Title: Virtual Reality Exercise During Hemodialysis
Brief Title: Virtual Reality During Hemodialysis
Acronym: VRHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital de Manises (Other); Universitat Politècnica de València (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/0638
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: End Stage Renal Disease; Hemodialysis-Induced Symptom
Keywords: exercise; physical function; health related quality of life
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants will receive during hemodialysis the conditions 'virtual reality exercise' for 12 weeks and 'control period-no exercise' for 12 more weeks
Who Masked: Investigator, Outcomes Assessor
Masking Description: A team of assessors, different to the researchers implementing the exercise, will record all dependent variables
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality during hemodialysis (Experimental): During 12 weeks subjects will exercise during hemodialysis. The intervention will be virtual reality exercise during hemodialysis.
  Interventions: Other: Virtual reality exercise during hemodialysis
- Control period - no exercise (No Intervention): During 12 weeks subjects will not exercise during hemodialysis

INTERVENTIONS:
Other: Virtual reality exercise during hemodialysis — Subjects will play a virtual reality game specially adapted for subjects undertaking hemodialysis treatment
  Arms: Virtual reality during hemodialysis

SUMMARY:
The main objective of this investigation is to assess if an intradialysis virtual reality exercise-based program results in an improvement in physical function and if it results in high adherence rates to exercise. The secondary aim is to assess the effect of intradialysis VR in physical activity level, health related quality of life and in cognitive function.

DETAILED DESCRIPTION:
Participants will be randomized into one of two groups. The first group will start with 12 weeks of virtual reality exercise during hemodialysis and will carry on with a control period of 12 weeks. The second group will start with a control period of 12 weeks (no exercise) and will carry on with a virtual reality exercise period of 12 weeks.

The virtual reality exercise will undertake up to 30 minutes of exercise. After warming up, participants will play to an adapted 'treasure hunt' game. Their legs movements will be the players projected into an individual tv that will give them feedback regarding their achievements. The aim of the game will be to achieve the higher possible score.They will move their legs to pick up coins and to avoid bombs. An adapted Kinect technology will be used for the game development. The exercise session will end-up with a cool-down period that will include simple lower limb stretching exercises.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months in hemodialysis treatment
* Clinically stable

Exclusion Criteria:

* Recent cardiac events (less than 3 months)
* Unable to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline gait speed at 12 weeks | Baseline, 12 weeks
  Speed to cover 4 meters at normal speed

SECONDARY OUTCOMES:
Change from baseline sit to stand 10 at 12 weeks | Baseline, 12 weeks
  Time to perform 10 sit to stand repetitions,
Change from baseline sit to stand 60 at 12 weeks | Baseline, 12 weeks
  Sit to stand repetitions performed in 60 seconds
Change from baseline timed up and go at 12 weeks | Baseline, 12 weeks
  Time to stand up, walk 3 meters, come back and sit down again
Change from baseline short physical performance battery at 12 weeks | Baseline, 12 weeks
  Score achieved at the battery that includes balance tests, sit to stand to sit 5 and and gait speed
Change from baseline handgrip at 12 weeks | Baseline, 12 weeks
  Bilateral handgrip strength
Change from baseline one-leg standing test at 12 weeks | Baseline, 12 weeks
  Time achieved while standing on one leg
Change from baseline one-leg heel rise test at 12 weeks | Baseline, 12 weeks
  Number of heel rise repetitions achieved
Change from baseline 6 minutes walk test at 12 weeks | Baseline, 12 weeks
  Number of meters walked in 6 minutes
Change from baseline Physical activity level at 12 weeks | Baseline, 12 weeks
  Physical activity questionnaires
Change from baseline Health related quality of life at 12 weeks | Baseline, 12 weeks
  Short Form 36 questionnaire to measure health-related quality of life
Change from baseline Cognitive function at 12 weeks | Baseline, 12 weeks
  Mini-mental State Examination questionnaire
Adherence | 12 weeks
  Sessions performed/sessions offered
Healthcare resources expenditure and costs | 12 months before starting the exercise program- 12 months after the starting date
  Total amount in euros spent on external consultations, laboratory tests, radiology tests, hospital pharmacy, emergency department healthcare provision, and hospitalisation.

CONTACTS AND LOCATIONS:
Overall Officials: Eva SEGURA-ORTÍ, PhD, Principal Investigator — Universidad CEU Cardenal Herrera, UCH CEU
Locations (1):
- Hospital de Manises, Manises, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Segura-Orti E, Gordon PL, Doyle JW, Johansen KL. Correlates of Physical Functioning and Performance Across the Spectrum of Kidney Function. Clin Nurs Res. 2018 Jun;27(5):579-596. doi: 10.1177/1054773816689282. Epub 2017 Jan 23. PMID 28114792
- [Background] Segura-Orti E, Martinez-Olmos FJ. Test-retest reliability and minimal detectable change scores for sit-to-stand-to-sit tests, the six-minute walk test, the one-leg heel-rise test, and handgrip strength in people undergoing hemodialysis. Phys Ther. 2011 Aug;91(8):1244-52. doi: 10.2522/ptj.20100141. Epub 2011 Jun 30. PMID 21719637
- [Background] Segura-Orti E, Johansen KL. Exercise in end-stage renal disease. Semin Dial. 2010 Jul-Aug;23(4):422-30. doi: 10.1111/j.1525-139X.2010.00766.x. PMID 20701722
- [Background] Segura-Orti E. [Exercise in haemodyalisis patients: a literature systematic review]. Nefrologia. 2010;30(2):236-46. doi: 10.3265/Nefrologia.pre2010.Jan.10229. Epub 2010 Jan 21. Spanish. PMID 20098466
- [Background] Segura-Orti E, Kouidi E, Lison JF. Effect of resistance exercise during hemodialysis on physical function and quality of life: randomized controlled trial. Clin Nephrol. 2009 May;71(5):527-37. doi: 10.5414/cnp71527. PMID 19473613
- [Background] Segura-Orti E, Rodilla-Alama V, Lison JF. [Physiotherapy during hemodialysis: results of a progressive resistance-training programme]. Nefrologia. 2008;28(1):67-72. Spanish. PMID 18336134